CLINICAL TRIAL: NCT04063878
Title: A Prospective, Multicenter Study on Acuris™ - Conometric Concept for Single Tooth Restoration. A 5-year Follow-up Study
Brief Title: A Clinical Study on Acuris™ - Conometric Concept for Single Tooth Restoration
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-OT-17-003
Record Dates: First submitted 2019-08-15; First posted 2019-08-21 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-02

CONDITIONS: Jaw, Edentulous, Partially
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single tooth restorations using Acuris conometric concept (Experimental)
  Interventions: Device: Conometric Abutment and Conometric Final Cap

INTERVENTIONS:
Device: Conometric Abutment and Conometric Final Cap — Conometric concept developed by Dentsply Sirona Implants for implant systems Ankylos, Astra Tech Implant System and Xive.

SUMMARY:
The purpose of this study is to evaluate the outcome of prosthetic survival of the Acuris conometric concept 1 year after permanent restoration, since this is a new mode of retention using friction for seating the crown of single tooth restorations without using cement or screws.

ELIGIBILITY:
Inclusion Criteria:

1. Subject aged between 18-75 years
2. Subject signed and dated the informed consent form
3. In need of an implant replacing a missing tooth in position 17 to 27 or 37 to 47, and each subject can only receive one study implant.
4. Neighbouring tooth to the planned implant must have

   * a natural root or an implant supported restoration mesially
   * a natural root or an implant supported restoration distally Exemption: If the planned implant is in the second molar position, an edentulous space is accepted distally.
5. Presence of natural tooth, partial prosthesis and/or implant supported restoration in the opposite jaw in contact with the planned crown
6. Deemed by the investigator as likely to present an initially stable implant situation

Exclusion Criteria:

1. Unlikely to be able to comply with study procedures, according to Investigators judgement
2. Subject is not willing to participate in the study or not able to understand the content of the study
3. Involvement in the planning and conduct of the study
4. Severe non-compliance to CIP as judged by the Investigator and/or Dentsply Sirona Implants.
5. Unable or unwilling to return for follow-up visits for a period of five years
6. Simultaneous participation in another clinical study, or former participation in a clinical study during the last 6 months that may interfere with the present study
7. Previous enrolment in the present study
8. Uncontrolled pathological process in the oral cavity
9. Known or suspected current malignancy
10. History of radiation therapy in the head and neck region within 12 months prior to surgery
11. Systemic or local disease or condition that could compromise post-operative healing and/or osseointegration
12. Uncontrolled diabetes mellitus
13. Corticosteroids, iv bisphosphonates or any other medication that could influence post-operative healing and/or osseointegration
14. Current need for major bone grafting and/or augmentation in the planned implant area (minor grafting and soft tissue grafting are allowed)
15. Smoking more than 10 cigarettes per day, present alcohol or drug abuse
16. Known pregnancy at implant installation (Only applicable for sites in United States and Canada)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2027-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Degidi, Dr., Principal Investigator — Degidi Dental Clinic, Bologna, Italy
Locations (9):
- United States (2):
  - University of Illinois College of Dentistry, Chicago, Illinois
  - Implant & Prosthodontic Associates, Oklahoma City, Oklahoma
- Cholakis Dental Group, Winnipeg, Canada
- Praxis Prof. Dr. Dhom & Kollegen MVZ GmbH, Ludwigshafen, Germany
- Studio Toia, Busto Arsizio, Italy
- Spain (2):
  - Clínica Dental Broseta, Cheste
  - Clinica Dental Antuña de Alaiz SL, Oviedo
- United Kingdom (2):
  - Ten Dental, London
  - The Implant Experts LTD, Maidstone

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Tooth Restorations Using Acuris Conometric Concept
Started | 160
Completed (1 year after permanent restoration) | 144 (Per protocol.)
Not Completed | 16
Not completed — Withdrawal by Subject | 2
Not completed — Subject not fulfilling study eligibility criteria | 14

BASELINE CHARACTERISTICS:
Arm/Group | Single Tooth Restorations Using Acuris Conometric Concept
Number analyzed (Participants) | 144
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.32 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 65
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Prosthetic Survival
Description: Evaluation of presence of original permanent restoration, remained retention between abutment and final cap, and occurrence of fracture/loss of abutment. Prosthetic survival will be categorized as No/Yes. It will be categorized as "Yes" if all of the following criteria are fulfilled:
  * Permanent restoration is remaining in situ.
  * No loss of conometric retention between abutment and final cap.
  * No fracture of abutment.
  * No loss of abutment.
Time Frame: 1 year after permanent restoration
Population: Per protocol 144 - Visit data missing for 13 participants.
Measure: Count of Units; unit: Permanent restorations
Units Other Than Participants: Permanent restorations
Arm/Group | Single Tooth Restorations Using Acuris Conometric Concept
Number analyzed (Participants) | 131
Number analyzed (Permanent restorations) | 131
Permanent restorations
  Prosthetic survival - Yes | 127
  Prosthetic survival - No | 4

2. Secondary Outcome: Prosthetic Survival
Time Frame: 3 and 5 years after permanent restoration
Reporting Status: Not Posted

3. Secondary Outcome: Implant Survival
Time Frame: 1, 3 and 5 years after permanent restoration
Reporting Status: Not Posted

4. Secondary Outcome: Marginal Bone Levels Alterations
Time Frame: 1, 3 and 5 years after permanent restoration
Reporting Status: Not Posted

5. Secondary Outcome: Bleeding on Probing
Description: Proportion of implants with any bleeding and proportion of bleeding surfaces
Time Frame: 1, 3 and 5 years after permanent restoration
Reporting Status: Not Posted

6. Secondary Outcome: Plaque
Description: Proportion of implants with any plack and proportion of all four surfaces with any plaque
Time Frame: 1, 3 and 5 years after permanent restoration
Reporting Status: Not Posted

7. Secondary Outcome: Probing Pocket Depth
Description: Measured aspects/side of implant; mean value, absolute value and changes.
Time Frame: 1, 3 and 5 years after permanent restoration
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From enrollment up to1 year after permanent restoration.
Arm/Group | Single Tooth Restorations Using Acuris Conometric Concept
All-Cause Mortality (participants affected / at risk) | 0/160
Serious Adverse Events (participants affected / at risk) | 4/160
Other Adverse Events (participants affected / at risk) | 8/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Tooth Restorations Using Acuris Conometric Concept (N=160)
COVID-19 (Infections and infestations) | 2 (2)
Renal colic (Renal and urinary disorders) | 1 (1)
Hypotensive crisis and renal insufficiency (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Tooth Restorations Using Acuris Conometric Concept (N=160)
Loss of conometric retention between abutment and final cap (Product Issues) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT04063878/Prot_SAP_000.pdf